CLINICAL TRIAL: NCT04620226
Title: Screening for Hepatitis C and Hepatitis B in Inpatients: A Toronto Viral Hepatitis Care Network (VIRCAN) Collaboration
Brief Title: UHN Inpatient Hepatitis C & B Screening
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Jordan Feld (Other)
Responsible Party: Sponsor-Investigator, Jordan Feld, Associate Professor, University Health Network, Toronto
Organization: University Health Network, Toronto (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: UHN Inpatient HCV & HBV Screen
Record Dates: First submitted 2020-10-01; First posted 2020-11-06 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Hepatitis C; Hepatitis B
Keywords: Hepatitis C; Hepatitis B; Screening; Inpatient; Hospital
MeSH Terms: conditions — Hepatitis C; Hepatitis B | interventions — Quality Improvement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Serum Testing (No Intervention): Participants will be screened by conventional HCV antibody (anti-HCV) serology and if screen positive, a second sample will be collected and tested for HCV RNA using a standard commercial assay.
- Rapid Point-of-Care Testing (Experimental): Participants will be screened using the OraQuick® Rapid Anti-HCV Point-of-Care Test (OraSure) and if screen positive, an additional whole blood sample will be collected and tested for HCV RNA using Xpert® HCV RNA (Cepheid) point-of-care testing and confirmed using a standard commercial assay.
  Interventions: Other: Quality Improvement

INTERVENTIONS:
Other: Quality Improvement — Rapid Point-of-Care testing will provide participants with a HCV antibody and RNA result within 2 hours. If the participant is HCV RNA+, they will receive an inpatient consultation from a liver specialist prior to discharge. We hypothesize that this model will minimize losses in the continuum-of-care and improve linkages to care.
  Arms: Rapid Point-of-Care Testing

SUMMARY:
Currently, there is a lack of literature on programs evaluating rapid screening methods to traditional venipuncture methods for sample collection during screening for viral hepatitis. Due to the relatively low diagnosis and linkage to care rate, screening programs that provide same day results for viral hepatitis infection may improve both diagnosis and enable providers to engage patients shortly after diagnosis. This stands in contrast to the multi-visit, weeks long process that normally accompanies serum testing for hepatitis C virus (HCV) and hepatitis B virus (HBV). A few American studies have examined the implementation of HCV inpatient screening programs; however, they are focused specifically on high-risk patient populations, the barriers to accessing care experienced by study participants are not relevant to the Canadian healthcare system context, and do not use rapid testing. Furthermore, there are few, if any, data on HBV inpatient screening programs and the diagnosis rate remains low. This project will provide key data on a rapid inpatient screening and linkage to care strategy as well as the prevalence of these viruses across different age bands within the population. Finally, the study will help determine whether rapid inpatient screening is a feasible and acceptable approach for screening and linkage to care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older at time of consent
* Patients admitted to GIMIUs at TGH or TWH

Exclusion Criteria:

* Patients whose end of life is expected to be less than 6 months
* Patients who are unable or decline to provide informed consent
* Patients with confirmed, active COVID-19 infections
* Patients with immediate life-threatening conditions where screening for chronic HCV and HBV infection may delay urgent care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2920 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Number of HCV antibody positive participants who complete an HCV RNA PCR. | 2 year
  To determine the proportion of HCV antibody positive participants who complete HCV RNA PCR in each arm. Participants will be contacted at 90 days and 1 year post-enrolment to self-report progress.
Number of HCV RNA positive participants who attend their first hepatology appointment. | 2 year
  To determine the proportion of HCV RNA positive participants successfully linked to care from each arm. Participants will be contacted at 90 days and 1 year post-enrolment to self-report.
Number of HCV RNA positive participants who achieve a Sustained Virological Response at 12 weeks (SVR12) after treatment completion. | 2 year
  To determine the proportion of HCV RNA positive participants who successfully achieved a sustained virological response at 12 weeks (SVR12) after treatment completion. Participants will be contacted at 90 days and 1 year post-enrolment to self-report.

SECONDARY OUTCOMES:
Number of chronic hepatitis C and hepatitis B infection in the general internal medicine inpatient units. | 1 year
  Proportion of screened participants who are positive and chronically infected in general internal medicine inpatient units.
Number of patients willing to participate in hepatitis C and hepatitis B screening in general internal medicine inpatient units. | 1 year
  To determine acceptability of implementing hepatitis C and hepatitis B screening in general internal medicine inpatient units.
Percentage of physicians, residents, and nurses who believe that hepatitis C and hepatitis B screening can be incorporated into the general internal medicine inpatient units' workflow. | 1 year
  To determine the effect of hepatitis C and hepatitis B screening on hospital staff workflow in general internal medicine inpatient units.
Proportion of Cepheid Xpert® HCV Viral Load test results matching test results from the standard commercial assay for HCV RNA PCR. | 1 year
  To determine whether results of the Cepheid Xpert® HCV Viral Load assay are valid when compared to the standard commercial assay for HCV RNA PCR.
Retrospective rates of HCV testing, HCV antibody positive results, and HCV RNA positive results in general internal medicine inpatient units. | 1 year
  To determine the historical rate of HCV screening and chronic HCV infection in general internal medicine inpatient units.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Toronto General Hospital, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No